CLINICAL TRIAL: NCT05721911
Title: Implementing a National Biobank of Genetic, Sporadic and Prodromic Parkinson's Disease With Whole Genome Analysis and Functional Assessment of Polygenic Inheritance by iPSC Technology
Brief Title: Implementing a National Biobank of PD With WGS and Functional Assessment of Polygenic Inheritance by iPSC Technology
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Neuromed IRCCS (Other)
Responsible Party: Principal Investigator, Teresa Esposito, Head of CNR Unit, Neuromed IRCCS
Other Study IDs: PNRR-MAD-2022-12375960
Record Dates: First submitted 2023-01-30; First posted 2023-02-10 (Actual); Last update posted 2023-02-15 (Actual); Status verified 2023-02

CONDITIONS: Parkinson Disease; REM Sleep Behavior Disorder
MeSH Terms: conditions — Parkinson Disease; REM Sleep Behavior Disorder | interventions — Whole Genome Sequencing

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples for purification of DNA, plasma and serum and PBMC. hiPSC will be generated by reprogramming of PBMC.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Genetic: whole genome sequencing — Partecipants will be assessed for disease progression: Stadio di Hoehn and Yahr, MDS-UPDRS part III, MOCA test, no motor symptoms, therapy and LID occurrence, Sleep disorders. Partecipants will be subjected to peripheral blood sampling for the purification of DNA, plasma, serum, PBMC and generation of hiPSC. DNA of each partecipants we will analysed by whole genome sequencing by next generation sequencing to identify any variant in candidate PD genes

SUMMARY:
The genetic complexity and heterogeneity of the sporadic forms of Parkinson's disease (PD) are posing a formidable challenge to disentangle their direct molecular causes. To advance this research, we plan to coordinate our local biorepositories of PD biological specimens creating a standardized and integrated national resource. In this framework, we plan to collect more samples from additional sporadic PD cases and to extend the sampling to patients with REM sleep behavior disease. We plan a large campaign of whole genome sequencing including about 200 patients to identify rare genomic variants plausibly associated with these diseases. In addition, we will standardize the generation and quality control of iPSC lines to make available to the scientific community. Finally, we will combine iPSC technology and gene editing to functionally assess the relative impact of rare variants in coding regions inherited together as a polygenic trait previously identified in selected sporadic PD cases

DETAILED DESCRIPTION:
The project is a multicentric observational study. Instuitutions involved are:

IRCCS Hospital San Raffaele, Milan Italy (coordinator Operating Unit (OU1)) IRCCS INM Neuromed, Pozzilli, (IS) Italy (Operating Unit (OU2)) IRCCS San Raffaele Roma, (Operating Unit (OU3)) The project takes advantage from the availability of a large collection of PD samples (~800) PD from familiar and sporadic cases, recruited at IRCCS Neuromed, for which we already collected and stored clinical information, genetic data as well as DNA, serum, plasma and peripheral blood mononuclear cells (PBMCs) for the entire study cohort.

The activities of the IRCCS INM Neuromed are:

1. standardization of the clinical reporting, sample collection, storage and identification between the centers;
2. recruitment of 100 PD patients, 30 RBD patients and 100 healthy subjects (patients' wives/husbands), to be carried out during the scheduled outpatient visits for these patients;
3. whole genome sequencing (WGS) and bioinformatic analysis (in collaboration with OU1) of a selected cohort of PD patients (200 samples), negative for mutations/variants in PD candidate genes;
4. WGS analysis of REM sleep behaviour disorder (RBD) prodromal patients as a model to identify early biomarker for PD;
5. development of an innovative protocol for early diagnosis of PD based on the co-inheritance of multiple rare deleterious variants in PD genes;
6. generation of induced pluripotent cell lines (iPSC) by reprogramming PBMCs from PD patients and familiar healthy donors.

After signed informed consent patients will be assessed for disease progression (Stadio di Hoehn and Yahr, MDS-UPDRS part III, MOCA test, no motor symptoms, therapy and LID occurrence, sleep behavior disease). Each patient and control will be subjected to peripheral blood sampling for the isolation of DNA, plasma, serum, PBMC. For a subset of patients induced pluripotent stem cells (iPSC) will be generated starting from PBMC.

Whole genome sequencing approach will be used to identify novel associated vatiants.

Extensive computational analysis will be planned to map the SNPs to regulatory regions controlling the expression of selected genes. This effort will provide the initial knowledge to draft the association between particular genomic SNPs and their combinations with sporadic PD. This endeavor is critical to advance our understanding of the genetic roots of PD and is in line with analogous ongoing international studies with whom will seek coordination. The success of this research will provide the means for developing predictive genetic testing and counselling of patients with PD and their families.

To increase the power analysis data will be analyzed including WES data of a cohort of 800 PD patients and 300 healthy subject already available at IRCCS INM Neuromed.

ELIGIBILITY:
Inclusion Criteria PD patients:

* Presence of at least 2 of the 4 cardinal signs (tremor, rigidity, bradykinesia, onset asymmetric) one of which must be tremor or bradykinesia;
* Absence of atypical symptoms such as: i) early postural instability, freezing phenomena, cognitive impairment, hallucinations, pathological involuntary movements, vertical gaze paralysis; ii) confirmed causes of secondary parkinsonism (focal lesions, drugs, substances toxic);
* Documented response to L-dopa or dopamine agonist use (or lack of adequate therapeutic attempt with L-dopa or dopamine agonists).

Inclusion Criteria RBD patients:

• Subjects affected by idiopathic RBD that will be selected according to the most recent criteria international classification of sleep disorders (ICSD-3).

Exclusion Criteria:

* pre-existing psychiatric conditions;
* Neurodegenerative neurological diseases such as multiple sclerosis, lateral sclerosis amyotrophic, Alzheimer's, neuromuscular pathologies, epilepsy;
* diagnosis of dementia;
* depression;
* prolonged intake of anxiolytics, antidepressants, antipsychotics, hypnotic drugs, cognitive stimulants

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study includes 100 PD patients, 30 RBD and 100 age/gender-matched controls. All PD patients will be diagnosed at the IRCCS Neuromed and followed-up (at least for 3 years) for disease progression
Sampling Method: Probability Sample
Enrollment: 230 (Estimated)
Dates: Start 2023-06 (Estimated); Primary Completion 2025-05 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
motor symptoms of PD and RBD patients will be evaluated with Hoehn and Yahr (HY) score | 2 years
  The Hoehn and Yahr Scale will be used to measure how Parkinson's symptoms progress and the level of disability. It includes stages 1 through 5: Stage 1. Unilateral involvement only, usually with minimal or no functional impairment; Stage 2 = Bilateral disease, without impairment of balance; Stage 3 = Mild to moderate bilateral disease; some postural instability; physically independent. Stage 4 = Severe disability; still able to walk or stand unassisted. Stage 5 = Wheelchair bound or bedridden unless aided.
motor and non motor symptoms of PD and RBD patients will be evaluated with MDS-UPDRS | 2 years
  The MDS-UPDRS has four parts, namely, I: Non-motor Experiences of Daily Living; II: Motor Experiences of Daily Living; III: Motor Examination; IV: Motor Complications. Twenty questions are completed by the patient/caregiver
clinical evaluation of of sleep disorders in PD and RBD patients | 2 years
  presence of sleep disorders will be evaluated by Munich Parasomnia Screening (MUPS)
clinical evaluation of of sleep disorders in PD and RBD patients by Polysomnography | 2 years
  Sleep microstructure will be evaluated by analysis of the alternating cyclic pattern (CAP), a marker of NREM sleep instability.
clinical evaluation of cognitive impairment of PD and RBD patients by MoCA test score | 2 years
  The Montreal Cognitive Assessment (MoCA) is a test used by healthcare providers to evaluate people with memory loss or other symptoms of cognitive decline. The MoCA contains 30 questions and checks different types of cognitive or thinking abilities. These include:orientation, short-term memory/delayed recall, executive function/visuospatial ability, clock-drawing test.
clinical evaluation of levodopa-induced dyskinesia (LID) in PD patients | 2 years
  LID occurrence will be related to levodopa dosage and time of therapy
identification of variants/mutations | 2 years
  the number of multiple rare (Minor allele frequency, MAF<0.01) deleterious (missense, non sense, frameshift and splicing) variants in PD genes will be counted in PD patients and unrelated healthy subjects. Case-control assoiciation study will evaluate the PD risk
association with phenotypic manifestation of PD | 2 years
  The presence of one or more variants will be tested for association with phenotypic manifestation of PD (motor, non motor, and cognitive signs, as well as age at onset, LID and neuroimaging changes) to assess the variant burden effect on progression, and prognosis of the disease

CONTACTS AND LOCATIONS:
Overall Officials: Teresa Esposito, PhD, Principal Investigator — IRCCS INM Neuromed
Locations (1):
- IRCCS Neuromed, Pozzilli, Italy

IPD SHARING:
Plan to Share IPD: Undecided
genetic data